CLINICAL TRIAL: NCT06686901
Title: A Randomized Controlled Trial of a Smartphone Delivered Treatment for Suicidal Thoughts and Behavior
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Adam C. Jaroszewski, PhD, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024P003049-phase2; K23MH133876 (NIH)
Record Dates: First submitted 2024-11-12; First posted 2024-11-13 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Suicidal Ideation; Suicide Attempt
Keywords: Suicide; ecological momentary assessment (EMA); Therapeutic Evaluative Conditioning (TEC)
MeSH Terms: conditions — Suicidal Ideation; Suicide, Attempted; Suicide

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Smartphone-delivered inactive Therapeutic Evaluative Conditioning (inactive TEC) (Placebo Comparator): Optional smartphone-delivered inactive Therapeutic Evaluative Conditioning (inactive TEC) for 30 days.
  Interventions: Behavioral: Smartphone-delivered inactive Therapeutic Evaluative Conditioning
- Smartphone-delivered active Therapeutic Evaluative Conditioning for Suicide (active TEC) (Experimental): Optional smartphone-delivered active Therapeutic Evaluative Conditioning for Suicide (active TEC-S) for 30 days.
  Interventions: Behavioral: Smartphone-delivered Therapeutic Evaluative Conditioning for Suicide (TEC-S)

INTERVENTIONS:
Behavioral: Smartphone-delivered Therapeutic Evaluative Conditioning for Suicide (TEC-S) — Therapeutic Evaluative Conditioning for Suicide (active TEC-S) is a behavioral treatment where participants are given optional access to a computerized task/game where they repeatedly pair suicidal behavior stimuli (pictures, words) with other negative stimuli and self-related stimuli with positive stimuli.
  Arms: Smartphone-delivered active Therapeutic Evaluative Conditioning for Suicide (active TEC)
Behavioral: Smartphone-delivered inactive Therapeutic Evaluative Conditioning — Therapeutic Evaluative Conditioning (inactive TEC-S) is a behavioral treatment where participants are given optional access to a computerized task/game where they repeatedly pair positive and negative stimuli (pictures, words) with each other.
  Arms: Smartphone-delivered inactive Therapeutic Evaluative Conditioning (inactive TEC)

SUMMARY:
This study aims to evaluate the acceptability, safety, and efficacy of a smartphone-delivered intervention called Therapeutic Evaluative Conditioning for Suicide (TEC-S) in reducing suicidal thoughts and behaviors (STB) among adults with recent and frequent suicide ideation.

DETAILED DESCRIPTION:
The present study is a two-arm randomized controlled trial (RCT) designed to evaluate the safety, acceptability, and efficacy of Therapeutic Evaluative Conditioning for Suicide (TEC-S), a smartphone-delivered intervention aimed at reducing suicidal thoughts and behaviors (STB). Participants in this study will be 60 adult participants (ages 18+) who report recent and frequent STB, residing within the greater-Boston, Ma area.

Participants will be randomized to receive either the control condition, which consists of 3x/daily ecological momentary assessment (EMA) of emotions and STBs and optional inactive TEC (n = 30), or the experimental condition, consisting of 3x/daily EMA and optional active TEC-S (n = 30). Evaluative conditioning uses classical conditioning to alter attitudes. The aim of TEC-S is to alter attitudes toward suicide and, in turn, reduce STB. EMAs will monitor STB, safety, and acceptability, and efficacy. Weekly behavioral and self-report assays will assess hypothesized treatment mechanisms. The study's aim is to determine if the active TEC-S condition reduces STB and to explore if altered attitudes toward suicide mediates this effect.

ELIGIBILITY:
Inclusion Criteria:

* Adults ages 18+
* Relatively frequent and recent (≥5 days within the past-month) active suicidal thoughts as assessed via SITBI-R.
* Willing and able to provide at least one emergency contact (name, phone number, relation).
* Owns an Android or iOS smartphone.
* Possesses at least occasional access to Wi-Fi-enabled internet for data down/uploads.
* Fluent in English and willing to provide informed consent.
* Living in the Boston metropolitan area (i.e., ~50 mile radius around Boston, MA)

Exclusion Criteria:

* Recent (past 3-month) hypo/manic symptoms or homicidal ideation or lifetime psychosis spectrum diagnosis as assessed via MINI 7.0.2.
* Recent acute suicide risk operationalized as affirmative responses to BOTH below items during structured clinical interview AND evaluation by the PI in consultation with Mentors/Advisor Drs. Wilhelm, Kleiman, and/or Bentley:
* At any time in past week: ≥ 8/10 current intent to act on suicidal thoughts (0 ["not at all"] to 10 ["extremely strong"]); AND
* At any time in past week: thought of a specific suicide plan (i.e, known method/means and/or location) with access to lethal means
* Impaired vision (e.g., legal blindness), technological illiteracy, or intellectual disability that might impair ability to provide valid data and/or informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2027-04-01 (Estimated); Primary Completion 2029-07-01 (Estimated); Study Completion 2029-08-31 (Estimated)

PRIMARY OUTCOMES:
Desire to die by suicide (Likert) | Through completion of treatment phase (day 1 through 30)
  Right now, how strongly do you want to kill yourself? [0 (not at all) to 10 (extremely)]; assessed via 3x/day ecological momentary assessment (Kleiman et al., 2018)

SECONDARY OUTCOMES:
Suicide intent (Likert) | Through completion of treatment phase (day 1 through 30)
  Right now, how strong is your intention to kill yourself today? [0 (I am definitely not going to kill myself today) to 10 (I am definitely going to kill myself today)]; assessed via 3x/day ecological momentary assessment
Suicide urge (Likert) | Through completion of treatment phase (day 1 through 30)
  Right now, how strong is your urge to kill yourself [0 (not at all) to 10 (very strong)]; assessed via 3x/day ecological momentary assessment.
Suicide thought incidence | Through treatment phase completed (day 1 through 30)
  Since the last survey, have you had suicidal thoughts? (yes/no); assessed daily via ecological momentary assessment
Suicide planning incidence | Through completion of treatment phase (day 1 through 30)
  Since the last survey, have you made a plan to kill yourself? (yes/no); assessed daily via ecological momentary assessment
Suicide preparation incidence | Through completion of treatment phase (day 1 through 30)
  Since the last survey, have you made any preparations to kill yourself? (yes/no); assessed daily via ecological momentary assessment.
Suicide attempt incidence | Through completion of treatment phase (day 1 through 30)
  Since the last survey, have you attempted to kill yourself? (yes/no); assessed daily via ecological momentary assessment
Suicidal behaviors (composite) | Through completion of treatment phase (day 1 through 30)
  A composite variable consisting of (i) suicide plan incidence, (ii) suicide preparation incidence, (iii) suicide attempt incidence, each assessed via ecological momentary assessment
Suicide aversion (AMP) | Through completion of treatment phase (day 1 through 30)
  Suicide aversion assessed implicitly/behaviorally via the Affect Misattribution Procedure (AMP; Payne et al., 2005)
Suicide aversion (Likert) | Through completion of treatment phase (day 1 through 30)
  Valence ratings of suicide-related pictures using a 9-point scale (-4 [extremely unpleasant] to 0 [neutral] to 4 [extremely pleasant]); assessed weekly (Jaroszewski et al., 2022).
Self affection (AMP) | Through completion of treatment phase (day 1 through 30)
  Self affection assessed implicitly/behaviorally via the Affect Misattribution Procedure (AMP; Payne et al., 2005)